CLINICAL TRIAL: NCT05712525
Title: Gut Recovery In Patients Following Surgery
Acronym: GRIPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: G-Tech Corporation (Industry)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CLP-2022-001
Record Dates: First submitted 2023-01-25; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Gastrointestinal Diseases; Ileus
MeSH Terms: conditions — Gastrointestinal Diseases; Ileus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: G-Tech Wireless Patch System (WPS) — Noninvasive monitoring of myoelectrical signals

SUMMARY:
The purpose of the study is to determine if the myoelectrical measurements made by the G-Tech Wireless Patch System correlate with clinical markers of postoperative recovery such as passage of flatus/bowel movement, oral tolerance of diet and discharge readiness. Subsequently the data will be studied to establish which information in the signals is important in determining when to feed patients and possibly discharge them..

DETAILED DESCRIPTION:
Measure myoelectric signals with the G-Tech WPS and determine if a correlation exists between signal strength and the rate of gastrointestinal recovery following surgery. Determine the relationship between gastrointestinal myoelectrical signal strength and clinical markers of recovery such as passage of flatus/bowel movement, oral tolerance of diet and discharge readiness.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to follow all study requirements
* Eighteen (18) years of age or older
* Subject is willing and able to follow all study requirements
* Subject will undergo a colectomy

Exclusion Criteria:

* Subject is pregnant or suspects pregnancy
* Known allergy to medical grade adhesive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo a colectomy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-10-07 (Actual); Primary Completion 2023-10-06 (Estimated); Study Completion 2024-10-06 (Estimated)

PRIMARY OUTCOMES:
GI Functional Recovery | 30 days after surgery
  Observe a correlation between signal strength and the rate of gastrointestinal recovery following surgery.

SECONDARY OUTCOMES:
Adverse Events | 30 days after surgery
  Anticipated adverse events through hospitalization; Unanticipated adverse events (UADEs) through hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Kristen Crowell, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States